CLINICAL TRIAL: NCT05709587
Title: Effects of Virtual Reality Training on the Balance, Gait, and Quality of Life Improvements of Patients With Stroke in the Subacute and Chronic Stages.
Brief Title: Impacts of Application of Virtual Reality on Gait and Balance for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20190135
Record Dates: First submitted 2023-01-11; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2020-01

CONDITIONS: Stroke
Keywords: stroke; balance; virtual reality; walking pace; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The subjects that received virtual reality functional gait training for 12 sessions. During the virtual reality intervention, they also received routine conventional rehabilitation therapy for twice a week, and training lasted for one hour. The 6-minute walking test (6MWT), 10-meter walk test (10MWT), Berg balance scale (BBS) and Chinese version of the Activities specific Balance Confidence scale were assessed pre- and post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality training group (Experimental): Virtual Reality training group: Three virtual environments employed in this study,time constraints,terrain changes, and moving obstacles were set to increase the difficulty of the walking task.The participants had to complete a task three times to proceed to the next level.
  Interventions: Other: Virtual reality training

INTERVENTIONS:
Other: Virtual reality training — Virtual reality Training for 12 sessions, two to three times for one week, one training session last for 20 minutes

SUMMARY:
The goal of this clinical trial is to learn about effects of virtual reality combined with conventional therapy on the balance, gait, and quality of life in stroke patients in the subacute and chronic stages. The main questions it aims to answer are:

• Virtual reality combined conventional therapy interventions can improve the gait, balance and functional status of stroke patients or not?

Participants will asked to do about 3 tasks in virtual reality intervention

* Walk in the flat ground
* Cross the obstacle on the ground
* Cross to moving obstacles

DETAILED DESCRIPTION:
The investigators referred to the scenes designed by previous studies to develop the three virtual environments employed in this study and made slight modifications according to Taiwan's conditions. Google Earth Virtual Reality (Google Inc., Mountain View, California, U.S., 2017) was uesd for the first and second task and Street Champ Virtual Reality (Zynk Software Srl , Cluj, Romania, 2016) was used for the third task.

Time constraints, terrain changes, and moving obstacles were set to increase the difficulty of the walking task. The speed obtained by the 10-m walking pretest was used as the training benchmark. The participants had to complete a task three times to proceed to the next level.

For Patient Registries: on-site audit.The subjects were referred from the rehabilitation Clinic of Kaohsiung Municipal Ta-Tung Hospital

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis of Stroke. 2. Must be able to ambulation with or without devices. 3. Were able to communicate and follow instructions. 4. Were rehabilitated at Kaohsiung Municipal Ta-Tung Hospital.

Exclusion Criteria:

* 1. Limb apraxia. 2. Any vision impairments. 3. Any hearing impairments. 4. Any vestibular impairments. 5. Any comorbidities that affected movements.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Walking pace | Measure changes from baseline walking pace tested before the intervention to one week after completion of all interventions.
  Use the 10 meters walking test to show the outcomes that presents in m/s.
Walking endurance | Measure changes from baseline walking distance tested before the intervention to one week after completion of all interventions.
  Use the 6 minutes walking test to show the outcomes that calculate the distance in meters.
Balance test | Measure changes from baseline Berg Balance Scale score tested before the intervention to one week after completion of all interventions.
  Use the Berg Balance Scale to show the balance outcomes. It consists of 14 items scored 0 to 4 for a total of 56 points. A higher score means lower fall risk.
Activities-specific balance confidence scale | Measure changes from baseline score of Chinese version of the activities-specific balance confidence scale tested before the intervention to one week after completion of all interventions.
  Use the Chinese version of the activities-specific balance confidence scale to show the outcomes.It consists of 15 items every item score on 0 to 100. 0 means no confidence to perform the tasks, 100 means fully confidence to finish tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chueh Tsai, BS, Principal Investigator — Kaohsiung Municipal Ta-Tung Hospital (Operation under entrustment with KMUH )
Locations (1):
- Kaohsiung Municipal Ta-Tung Hospital (operation under entrustment with Kaohsiung Medical University Hospital), Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fung J, Richards CL, Malouin F, McFadyen BJ, Lamontagne A. A treadmill and motion coupled virtual reality system for gait training post-stroke. Cyberpsychol Behav. 2006 Apr;9(2):157-62. doi: 10.1089/cpb.2006.9.157. PMID 16640470
- [Background] Richards CL, Malouin F, Lamontagne A, McFadyen BJ, Dumas F, Comeau F, Robitaille NM, Fung J. Gait Training after Stroke on a Self-Paced Treadmill with and without Virtual Environment Scenarios: A Proof-of-Principle Study. Physiother Can. 2018 Summer;70(3):221-230. doi: 10.3138/ptc.2016-97. PMID 30275647